CLINICAL TRIAL: NCT03140592
Title: EUS-guided Biopsy of Pancreatic Mass Lesions for Developing Patient -Derived Cancer Models
Brief Title: Pancreatic Cancer Models Developed From EUS Guided Biopsy Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jonathan Buscaglia, Associate Professor, Stony Brook University
Other Study IDs: IRBNet # 618834
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma; Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsies of your pancreatic mass
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsy — Two extra EUS guided pancreatic biopsies collected for only research purposes.

SUMMARY:
Pancreatic cancer is a very aggressive cancer. Over the past 40 years there has not been much progress made in reducing deaths from this cancer. Recently, new models of pancreatic cancers have been generated from mouse and human tissues. These models have used larger pieces of tissues taken from surgical removal of pancreatic cancers.

The purpose of this study is to determine whether these new pancreatic cancer models can be generated from the small biopsies we take to make the diagnosis of the pancreatic mass.

DETAILED DESCRIPTION:
The Endoscopic Ultrasound guided pancreatic biopsy tissue collected for only research purposes will be used to generate organoids in a in-vivo and in-vitro setting.

The development of these methods may help scientists identify new treatments for pancreatic cancer and to potentially develop more personalized approaches to treating pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for an EUS-FNB of pancreatic mass(es) suspicious for pancreatic ductal adenocarcinoma performed by a member of the Stony Brook Interventional Endoscopy Section of the Division of Gastroenterology and Hepatology

1. Age ≥ 18 years
2. Literate and able/willing to provide informed consent for participation in research.

Exclusion Criteria:

1. Age < 18 years
2. Not literate or unable/unwilling to provide informed consent for EUS-FNB research biopsies
3. Pregnancy as determined by serum or urine HCG test performed as standard of clinical care for all women of childbearing age and documented on subjects' electronic medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for an EUS-FNB performed by a member of the Stony Brook Interventional Endoscopy Section of the Division of Gastroenterology and Hepatology
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01-14 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Successful generation of pancreatic organoids | 6 years
  The two extra biopsy tissues collected for only research purposes will be used to generate pancreatic organoids in a in-vivo as well as in-vitro setting.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Buscaglia, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacomb JF, Plenker D, Tiriac H, Bucobo JC, D'souza LS, Khokhar AS, Patel H, Channer B, Joseph D, Wu M, Tuveson DA, Li E, Buscaglia JM. Single-Pass vs 2-Pass Endoscopic Ultrasound-Guided Fine-Needle Biopsy Sample Collection for Creation of Pancreatic Adenocarcinoma Organoids. Clin Gastroenterol Hepatol. 2021 Apr;19(4):845-847. doi: 10.1016/j.cgh.2020.02.045. Epub 2020 Feb 29. PMID 32119924
- [Derived] Tiriac H, Bucobo JC, Tzimas D, Grewel S, Lacomb JF, Rowehl LM, Nagula S, Wu M, Kim J, Sasson A, Vignesh S, Martello L, Munoz-Sagastibelza M, Somma J, Tuveson DA, Li E, Buscaglia JM. Successful creation of pancreatic cancer organoids by means of EUS-guided fine-needle biopsy sampling for personalized cancer treatment. Gastrointest Endosc. 2018 Jun;87(6):1474-1480. doi: 10.1016/j.gie.2017.12.032. Epub 2018 Jan 9. PMID 29325707